CLINICAL TRIAL: NCT00366782
Title: A Phase 1 Study of the Safety and Immunogenicity of the Recombinant Live-Attenuated Chimeric Bovine/Human Parainfluenza Type 3 Virus Vaccine, rB/HPIV3, Lot PIV3 #101A, Delivered as Nose Drops to Adults 18 to 49 Years of Age, HPIV3-Seropositive Children 15 to 59 Months of Age, and HPIV3-Seronegative Infants and Children 6 to 36 Months of Age
Brief Title: Safety of and Immune Response to a Cow/Human Parainfluenza Virus Vaccine (rB/HPIV3) in Healthy Infants, Children, and Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 231; WIRB Protocol Number 20061455
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Paramyxoviridae Infections; Virus Diseases
Keywords: Respiratory Tract Disease; Bovine; Chimeric Vaccine
MeSH Terms: conditions — Paramyxoviridae Infections; Virus Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): One vaccination with rB/HPIV3 vaccine (at higher dose) given as nose drops to adults 18 to 49 years of age
  Interventions: Biological: rB/HPIV3
- 2 (Experimental): One vaccination with rB/HPIV3 vaccine (at higher dose) given as nose drops to HPIV3-seropositive children 15 to 59 months of age). This arm may enroll after Arm 1 depending on the effect of the vaccine on Arm 1.
  Interventions: Biological: rB/HPIV3
- 3 (Experimental): One vaccination with rB/HPIV3 vaccine (at lower dose) given as nose drops to seronegative children or infants 6 to 36 months of age. This arm may enroll after Arm 2.
  Interventions: Biological: rB/HPIV3
- 4 (Experimental): One vaccination with rB/HPIV3 vaccine (at higher dose) given as nose drops to seronegative children or infants 6 to 36 months of age. This arm may enroll after Arm 2.
  Interventions: Biological: rB/HPIV3
- 5 (Placebo Comparator): One vaccination with placebo vaccine given as nose drops to adults, HPIV3-seropositive children, or seronegative children or infants
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rB/HPIV3 — Live attenuated rB/HPIV3 vaccine given at a dose of 10^6 TCID50
  Arms: 1; 2; 4
Biological: rB/HPIV3 — Live attenuated rB/HPIV3 vaccine given at a dose of 10^5 TCID50
  Arms: 3
Biological: Placebo — Placebo for rB/HPIV3 vaccine
  Arms: 5

SUMMARY:
Human parainfluenza viruses (HPIVs) are a major health concern in infants and young children under 5 years of age, causing serious respiratory tract disease. The purpose of this study is to test the safety of and immune response to a new HPIV vaccine in healthy infants, children, and adults.

DETAILED DESCRIPTION:
HPIV type 3 (HPIV3) ranks second only to respiratory syncytial virus as the most common cause of bronchiolitis and pneumonia in infants less than 6 months of age. HPIV3 can cause severe disease in the first 2 years of life and is responsible for 11% of hospitalizations for respiratory diseases in children. This study will evaluate the safety and immunogenicity of a live, chimeric bovine/human, attenuated intranasal HPIV3 vaccine, rB/HPIV3. This vaccine combines modified human HPIV3 with a related, modified cow virus, bovine parainfluenza type 3 virus (BPIV3). Vaccinations will be given as nose drops to healthy adults, children seropositive for HPIV3, and infants and children seronegative for HPIV3.

There are four groups in this study. Group 1 will consist of adults who will receive the higher dose of rB/HPIV3. Group 2 will consist of seropositive children who will be randomly assigned to receive the higher dose of rB/HPIV3 or placebo. Group 2 will not begin enrollment until the completion of Group 1 safety data review. Participants of both Groups 1 and 2 will be monitored for 10 days post vaccination for respiratory illness and for fever by self-reported temperature logs; these participants will be followed for a maximum of 28 days. Blood collection will occur at study entry and on Day 28; additional blood collection may occur up to 28 days prior to vaccination. Clinical assessments and nasal washes will occur at study entry and selected study visits. Group 1 participants will be contacted by phone on Day 180; Group 2 participants' parents or guardians will be contacted by phone on Days 1, 2, 8, 9, 11, and 180; study staff will ask about any illnesses or adverse events that may have occurred.

Groups 3 and 4 will consist of seronegative infants and children. Group 3 will not begin enrollment until the completion of Group 2 safety data review. Children in Group 3 will be randomly assigned to receive the lower dose of rB/HPIV3 or placebo. Group 4 will not begin enrollment until the completion of Group 3 safety data review. Children in Group 4 will be randomly assigned to receive the higher dose of rB/HPIV3 or placebo. Participants of both Groups 3 and 4 will be monitored closely for 28 days postvaccination for respiratory illness and for fever by self-reported temperature logs; these participants will be followed for a maximum of 56 days. Blood collection will occur at study entry and on Day 56. Clinical assessments and nasal washes will occur at study entry and most study visits. Participants' parents or guardians will be contacted by phone periodically post vaccination; study staff will ask about any illnesses or adverse events they may have observed in their infants or children.

ELIGIBILITY:
Inclusion Criteria for Adult Participants:

* Good general health
* Available for the duration of the trial
* Reachable by telephone for post-vaccination contact
* Female participants willing to use acceptable methods of contraception

Inclusion Criteria for Seropositive Child Participants:

* Good general health and age-appropriate development, as determined by physical exam and medical history review
* Seropositive for human parainfluenza type 3 virus (HPIV3), as defined by a serum hemagglutination-inhibition (HI) antibody titer of more than 1:8
* Available for the duration of the trial
* Parent or guardian willing to provide informed consent
* Parent or guardian reachable by telephone for post-vaccination contact

Inclusion Criteria for Seronegative Infant and Child Participants:

* Good general health and age-appropriate development, as determined by physical exam and medical history review
* Seronegative for HPIV3, as defined by serum HI antibody titer of 1:8 or less within 28 days of first vaccination
* Available for the duration of the trial
* Parent or guardian willing to provide informed consent
* Parent or guardian reachable by telephone for post-vaccination contact

Exclusion Criteria for Adult Participants:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the participant to understand and cooperate with the study
* Medical, work-related, or family problems as a result of alcohol or illicit drug use in the 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Absence of spleen
* Diagnosis of asthma within the 2 years prior to study entry
* HIV-1 infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Abnormal blood or urine tests
* Known immunodeficiency syndrome
* Blood products, including immunoglobulin, within the 3 months prior to study entry
* Immune globulin within 3 months of vaccination
* Current smoker unwilling to stop smoking for the duration of the study
* Participation in another investigational vaccine or drug trial within 30 days of vaccination or while participating in this study
* Live vaccine within 4 weeks of vaccination
* Killed vaccine within 2 weeks of vaccination
* Previous immunization with PIV3 vaccine
* Known hypersensitivity to any vaccine component
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Work and/or personal responsibilities that involve caring for children less than 6 months of age or immunosuppressed individuals
* Pregnancy or breastfeeding

Exclusion Criteria for Infant and All Child Participants:

* Known or suspected impairment of immune system, including maternal history of positive HIV test, previous receipt of immunosuppressive therapy including systemic corticosteroids, or receipt of bone marrow/solid organ. Participants who have received topical steroids are not excluded.
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with PIV3 vaccine
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Lung or heart disease, including reactive airway disease. Participants with clinically insignificant cardiac abnormalities not requiring treatment are not excluded. More information on this criterion can be found in the protocol.
* Clinically significant abnormality in liver function test (seropositive participants only)
* Clinically significant abnormality in complete blood count (CBC) (seronegative participants only)
* Member of a household that includes a pregnant woman, an immunocompromised individual, or an infant less than 6 months of age
* Attends day care with infants less than 6 months of age, pregnant caregivers, or immunosuppressed individuals
* Parent or guardian unwilling to suspend day care for 14 days following vaccination. More information on this criterion can be found in the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of first vaccination or while participating in this study

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2007-03; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events (REs) that occur during the acute monitoring phase of the study (Days 0 to 10 for adult and seropositive groups, Days 0 to 28 for seronegative groups) | Throughout study
Quantifying the amount of vaccine virus shed by each recipient | Throughout study
Determining the amount of serum antibody and mucosal antibody induced by the vaccine in each recipient | Throughout study

SECONDARY OUTCOMES:
Determining the phenotypic stability of vaccine virus shed | Throughout study
Determining the number of vaccinated children and infants infected with rB/HPIV3 vaccine virus | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Durbin AP, Karron RA. Progress in the development of respiratory syncytial virus and parainfluenza virus vaccines. Clin Infect Dis. 2003 Dec 15;37(12):1668-77. doi: 10.1086/379775. Epub 2003 Nov 20. PMID 14689350
- [Background] Greenberg DP, Walker RE, Lee MS, Reisinger KS, Ward JI, Yogev R, Blatter MM, Yeh SH, Karron RA, Sangli C, Eubank L, Coelingh KL, Cordova JM, August MJ, Mehta HB, Chen W, Mendelman PM. A bovine parainfluenza virus type 3 vaccine is safe and immunogenic in early infancy. J Infect Dis. 2005 Apr 1;191(7):1116-22. doi: 10.1086/428092. Epub 2005 Feb 22. PMID 15747247
- [Background] Lee MS, Greenberg DP, Yeh SH, Yogev R, Reisinger KS, Ward JI, Blatter MM, Cho I, Holmes SJ, Cordova JM, August MJ, Chen W, Mehta HB, Coelingh KL, Mendelman PM. Antibody responses to bovine parainfluenza virus type 3 (PIV3) vaccination and human PIV3 infection in young infants. J Infect Dis. 2001 Oct 1;184(7):909-13. doi: 10.1086/323150. Epub 2001 Aug 15. PMID 11509996
- [Background] Madhi SA, Cutland C, Zhu Y, Hackell JG, Newman F, Blackburn N, Murphy BR, Belshe RB, Karron RA, Deatly AM, Gruber WC, Bernstein DI, Wright PF. Transmissibility, infectivity and immunogenicity of a live human parainfluenza type 3 virus vaccine (HPIV3cp45) among susceptible infants and toddlers. Vaccine. 2006 Mar 20;24(13):2432-9. doi: 10.1016/j.vaccine.2005.12.002. Epub 2005 Dec 20. PMID 16406170
- [Result] Karron RA, Thumar B, Schappell E, Surman S, Murphy BR, Collins PL, Schmidt AC. Evaluation of two chimeric bovine-human parainfluenza virus type 3 vaccines in infants and young children. Vaccine. 2012 Jun 6;30(26):3975-81. doi: 10.1016/j.vaccine.2011.12.022. Epub 2011 Dec 14. PMID 22178099